CLINICAL TRIAL: NCT05184023
Title: A Double-Blinded, Randomized-Controlled-Trial to Investigate the Effect of Pulsed Electromagnetic Field (PEMF) for Patients With Quadriceps Weakness After Anterior Cruciate Ligament Reconstruction (ACLR)
Brief Title: The Effect of PEMF for Patients With Quadriceps Muscle Weakness After ACLR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021.332
Record Dates: First submitted 2021-11-23; First posted 2022-01-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Anterior Cruciate Ligament Injuries; Quadriceps Muscle Atrophy
Keywords: Pulsed electromagnetic field; PEMF; Quadricep Strength; ACL; ACLR
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into either treatment group or sham group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: It is doubled blinded, a subject 's specific ID card will be provided for each of the enrolled subject and the investigators don't know whether it is PEMF or Sham treatment for that subject's specific ID card. And the investigator will ask the manufactory about the number of grouping at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Device: Pulse Electromagnetic Field
- Sham group (Sham Comparator)
  Interventions: Device: Sham Pulse Electromagnetic Field

INTERVENTIONS:
Device: Pulse Electromagnetic Field — Subjects will receive PEMF treatment with the duration of 8 weeks, twice a week with total 16 treatment sessions.
  Arms: Treatment group
Device: Sham Pulse Electromagnetic Field — Subjects will receive sham PEMF treatment with the duration of 8 weeks, twice a week with total 16 treatment sessions.
  Arms: Sham group

SUMMARY:
In Hong Kong, over 3000 Anterior Cruciate Ligament Reconstructions (ACLR) are performed each year in order to restore knee function after an ACL injury. The ultimate goal of ACLR is to fulfil the return-to-play (RTP) criteria. Despite successful surgery and a demanding rehabilitation process, some athletes still fail to comply to RTP. For those who achieve RTP, 23% of those who return to their sports would suffer a second ACL injury.

Quadriceps muscle strength is one of the key determinants for a patient's successful return- to-play after ACLR. Quadriceps muscle atrophy can persist beyond the completion of the rehabilitation program in almost half the patients and the reason behind this is still unknown. Therefore, there is need to find a more effective way to increase quadriceps strength.

There are emerging evidences showing that pulsed electromagnetic field (PEMF) can modulate mitochondrial activities for muscle gain. PEMF exposure on top of regular exercise training may promote muscle regeneration and tissue healing.

This study aims to conduct a double-blinded, randomized controlled trial to investigate the effects of PEMF treatment during the late postoperative period on quadriceps muscle strength in ACL injured patient. Muscle endurance could only be investigated in late postoperative period. The investigators hypothesize that PEMF treatment is effective to reduce muscle weakness and promote gain in quadriceps muscle strength in ACLR patients.

Based on the aim of this study, adult patients (aged 18-30) with a unilateral ACL injury, total quadriceps muscle volume is equal or morn than 7% deficit on involved leg compared with uninvolved leg, sporting injury with a Tegner score of 7+, both knees without a history of injury/prior surgery will be recruited. To estimate the improvement of patients, Isokinetic muscle assessment, ultrasound imaging and MRI for quadriceps muscle thickness, self-reported outcomes with questionnaires, KT-1000 for knee laxity and biomechanical analysis, Xtreme CT for Bone mineral density will be performed.

To investigate the mechanism of PEMF therapy on increasing quadriceps strength, samples of blood serum will be draw before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 with a unilateral ACL injury
2. Sporting injury with a Tegner score of 7+
3. LSI for quadriceps strength <70% of the contralateral leg at 4 months post-up
4. Both knees without a history of injury/prior surgery

Exclusion Criteria:

1. Ages smaller than 18 years old or greater than 50 years old
2. Any concomitant bone fracture, major meniscus injury or full-thickness chondral injuries requiring altered rehabilitation program post-op
3. Preoperative radiographic signs of arthritis
4. Metal implants that would cause interference on MRI
5. Non-HS graft for ACLR
6. Patient non-compliance to the rehabilitation program
7. Pregnancy or possibility of pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of peak torque of Isokinetic muscle strength | pre intervention, 4weeks, 8 weeks and 8 months after the commencement of intervention
  The peak torque in N will be the single highest repetition value within the 30 repetitions in the isokinetic muscle strength test.
Change of Fatigue index of isokinetic muscle strength | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The Fatigue index (F.I) can be used to calculated the percent decrease for each variable which reflected the muscle endurance.

SECONDARY OUTCOMES:
MRI Muscle thickness | pre PEMF intervention and 8 weeks after the commencement of intervention
  Muscle volumes of quadriceps muscle are measured using a 1.5 or 3.0 Tesla MRI Scanner. Axial (3mm thick cut) T1W images are obtained from the anterior superior iliac spine (ASIS) to the patella. Quadriceps muscles were manually outlined in each axial slice. Muscle volume was calculated by summing all of the slice-multiplied by slice thickness. The quality of the muscle is assessed by analyzing the fat content of the muscle mass using a technique that has been reported by Reeder et al. Scans will be performed on both legs before the start of the PEMF treatment (4 months post-op) and only on the injured side repeated after the completion of the 8 weeks PEMF treatment (6 months post-op). The uninjured side will be used as a reference for 'normal volume'.
Ultrasound imaging muscle thickness | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The Aixplorer® ultrasound system and a linear transducer probe with a bandwidth of 2-10 MHz were used to measure the muscle thickness of Vastus Medialis (VM), Vastus Lateralis (VL), and Rectus Femoris (RF) on both the injured and uninjured leg. Participants laid supine on a treatment table for the assessment. A measuring tape was used to locate VM, VL, RF and the patella by palpation, consequently marked with a pen for reference. RF was marked at 1/2 of the distance from the anterior superior iliac spine (ASIS) to the superior pole of the patella, VM was located at 1/5 of the distance away from the midpoint of the medial patella border to the ASIS, and VL was noted at 1/3 of the distance from the midpoint of the lateral patella border to the ASIS. After locating the anatomical points, excess contact gel was applied on these points. The transducer probe was aligned in the transverse plane and moved along the entire muscle bundle to capture a view of the VM, VL and RF.
Serum myokine evaluation | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  Phlebotomy (5ml) will be performed on the day before PEMF treatment, at 4- and 8- weeks after commencement of treatment, and at 8 months after the commencement of intervention. The serum will be prepared by centrifugation and kept in a -80o freezer until use. Quantitative analysis for myokines and proteins related to muscle metabolism will be performed by Human Myokine Magnetic Bead Panel (Millipore) with Bioplex-200 bead-based suspension assay system (LKSIHS core facilities), or enzyme-linked immunosorbent assay (ELISA) and report with pg/ml. These include Brain-derived neurotrophic factor (BDNF), Fibroblast growth factor-21 (FGF-21), Interleukin-6 (IL-6), IL-15, Irisin, Myostatin (MSTN)/GDF8, Insulin-like growth factor 1 (IGF-1), FGF-2, IL-8, Follistatin, Musclin, Myonectin, Decorin, Meteorinlike, Osteopontin, Secreted protein acidic and rich in cysteine (SPARC), Klotho, Procollagen type III N-terminal peptide (P3NP), and C- terminal of troponin T1 (TNNT1).
Passive Knee laxity | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  To measure anterior-posterior knee laxity, the KT-1000 knee ligament arthrometer (MEDmetric Corp, San Diego, CA, USA) will be used. A manual force test will be applied until a 30lb sound signal is activated. Three trials will be performed. A side difference of 3 mm above is considered clinically relevant.
Reaming size of the bone | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The reaming size of the bone in mm on the involved side will be scanned by XtremeCT II which provides an analysis of bone microarchitecture at human peripheral sites with high spatial resolution and low exposure to radiation.
Ground reaction force | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The Kinetic variables including vertical and horizontal ground reaction force (GRF) will be evaluated by a synchronized force plate at the centre of the capture volume at 1000Hz.
Knee Joint moments | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  The kinematics will be assessed by the skin marker-based motion analysis system with the lower-body marker setup followed the OSTRC standard using 16-camera and 16 reflective skin marker during the single leg squat and single leg hop test.
Single leg hop distance | 4weeks, 8 weeks and 8 months after the commencement of intervention
  The average of single leg hop distance in cm with three attempts will be measured during the single leg hop test.
Visual Analogue Scale | Before and after 1st - 16th of PEMF treatment
  The subjective measurement for chronic and acute pain will be recorded by the Visual Analogue Scale (VAS). VAS consists of a 10-cm line which represents the continuum between "painless" and "worst pain from 0 cm to 10 cm. The subject will be asked to draw a mark of it before and after each PEMF treatment session.
Tegner activity score | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  This is an activity level scaled from 1 (low activity) to 10 (high activity).
International Knee Documentation Committee | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  Consists of 10 questions on symptoms and activity ranging from 0 to 100 where 100 implies perfect knee function.
Lysholm knee scoring system | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  Consists of eight items, total score ranging from 0 to 100 where higher scores indicate a better outcome with fewer symptoms or disability.
International Physical Activity Questionnaire | pre PEMF treatment , 4weeks, 8 weeks and 8 months after the commencement of intervention
  Consists of four items recording the subject's time of spending on physical activities during the past 7 days with a validated Chinese version of the quantitative physical activity questionnaire, and the physical activity level will be evaluated by Metabolic Equivalent of task(MET) per minute and classified as physical level with Low, Moderate or High.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tim-Yun Ong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewers

REFERENCES:
- [Derived] Ong MT, Man GC, Lau LC, He X, Qiu J, Wang Q, Chow MC, Choi BC, Yu M, Yung PS. Effect of pulsed electromagnetic field as an intervention for patients with quadriceps weakness after anterior cruciate ligament reconstruction: a double-blinded, randomized-controlled trial. Trials. 2022 Sep 12;23(1):771. doi: 10.1186/s13063-022-06674-2. PMID 36096886

DOCUMENTS (2):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT05184023/Prot_000.pdf
  • Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT05184023/ICF_001.pdf